CLINICAL TRIAL: NCT02383160
Title: A Randomized Controlled Trial Comparing Low-Intensity, Pulsed Ultrasound to Placebo in the Treatment of Operatively Managed Scaphoid Non-Unions
Brief Title: Scaphoid Non-union and Low-intensity Pulsed Ultrasound Trial
Acronym: SNAPU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Workers' Compensation Board, Alberta (Other); Calgary Orthopaedic Research and Education Fund (Other); Bioventus LLC (Industry)
Responsible Party: Principal Investigator, Neil White, Clinical Assistant Professor, Section of Orthopaedics, Hand & Wrist Surgeon, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB13-0849
Record Dates: First submitted 2015-02-26; First posted 2015-03-09 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Nonunion of Fracture of Scaphoid Bone; Fractures, Ununited
Keywords: Low-intensity pulsed ultrasound; Nonunion; Scaphoid; Operative
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active LIPUS Unit (Active Comparator): Low-intensity pulsed ultrasound treatment 20 minutes/day until the fracture is deemed united clinically and on CT scan.
  Interventions: Device: Bioventus Exogen 4000: Low-intensity pulsed ultrasound
- Sham LIPUS Unit (Sham Comparator): Sham device treatment 20 minutes/day until the fracture is deemed united clinically and on CT scan.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Bioventus Exogen 4000: Low-intensity pulsed ultrasound — Active low-intensity pulsed ultrasound
  Other Names: Bioventus Exogen 4000
  Arms: Active LIPUS Unit
Device: Sham device — Placebo device with no active therapy
  Other Names: Bioventus Exogen 4000 Sham Unit
  Arms: Sham LIPUS Unit

SUMMARY:
This is a prospective, double-blind, multicentered, randomized controlled trial to determine the effectiveness of low-intensity pulsed ultrasound in decreasing the time to union of scaphoid non-unions after operative fixation as measured by serial CT scanning. Multiple centers across Canada will be involved in the study. Blinding will include patients, surgeons, research assistants, as well as all data handlers and analysts until trial completion or mid-term analysis.

DETAILED DESCRIPTION:
This is a prospective, double-blind, multicentered, randomized controlled trial to determine the effectiveness of low-intensity pulsed ultrasound in decreasing the time to union of scaphoid non-unions after operative fixation as measured by serial CT scanning. Multiple centers across Canada will be involved in the study. Blinding will include patients, surgeons, research assistants, as well as all data handlers and analysts until trial completion or mid-term analysis. Baseline demographics including age, hand dominance, work status and medical co-morbidities of the patients will be collected to allow for comparison of the groups to ensure similarity.

Patients will be identified during clinic appointment for the initial consultation for surgical fixation of their scaphoid non-union. Patients consenting to surgical fixation will be assessed for inclusion and exclusion criteria and, if appropriate, will be consented and evaluated for baseline range of motion, grip strength, SF-36, DASH and both resting and activity VAS scores. Pre-operative radiographs will be assessed for the degree of wrist arthritis present. No restrictions will be placed on the selection or scheduling of surgical procedures, but the use of other adjuvants such as bone morphogenic protein will be limited.

Bioventus will provide visually identical active and sham Exogen 4000 units. The units will undergo randomization and will be given consecutively numbered labels. Devices will be securely stored at each clinical study center. All clinical centers and personnel involved will be blinded to the randomization. Two weeks post-operatively subjects will attend the cast clinics and be assigned the next sequential device. The device will be applied through a window cut into the standardized cast with a center point over the anatomic snuffbox. This cast will remain in place until the fracture is united on CT or 7 weeks at a minimum.

Treatment will be self-administered for 20 minutes once daily by the patients. The device will be equipped with a system to document compliance with the treatment. Treatment will continue until the subject has greater than 50% cortical bridging on CT scanning with multi-planar reconstruction. Union will be confirmed by both an orthopedic surgeon and an independent musculoskeletal radiologist. Treatment will also be terminated if the subject continues to have non-union present at 6 months postoperatively. Subjects will be assessed for trabecular bridging using serial CT scans until the union is documented. CT scans will take place every 4-6 weeks until union is established. Standard scaphoid and wrist radiographs will be completed within 1 week of the CT scan. Patients who do not have documented union will be classified as persistent non-unions but will be asked to continue and attend clinical follow-ups until 1 year. Patients will be required to attend follow up visits at 2, 8, 12, 16, 24, 52 and 104 weeks for functional assessments. Patients requiring additional surgery such as bone grafting as deemed necessary by their treating surgeon will be scheduled at the surgeon's discretion and the surgery will be recorded as a trial adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a scaphoid fracture > 3 months-old with at least one feature of non-union including, collapse or humpback deformity, sclerosis at the fracture site or cystic changes evident on pre-operative diagnostic imaging
* Subject has consented to surgical fixation at surgeon discretion
* Subject is willing and has the ability to operate the LIPUS device for at least four to six months post-operatively

Exclusion Criteria:

* Subject with concomitant fracture or dislocation of another ipsilateral carpal bone, distal radius or ulna, or bilateral scaphoid fractures
* Subject has an open or pathological fracture
* Subject who are actively receiving treatment of a rheumatologic disorder with a biologic medication or other arthritic condition
* Subject has a history of fibrous dysplasia, chronic renal failure, Paget's disease, osteopetrosis or other impairing disease/condition of the musculoskeletal system
* Subject with an active infection of the affected limb
* Subject with a high risk of death within the follow up period
* Subject is a prisoner or at high risk of incarceration
* Subject who are unlikely to complete follow-up (no fixed address, states they are unlikely to complete follow up, psychiatric condition at surgeon discretion)
* Subject has cognitive impairment or language difficulties that would impede the completion of questionnaires
* Subject who are pregnant or anticipate getting pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2014-09; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to radiographic union as evidenced on serial CT scans | up to 52 weeks

SECONDARY OUTCOMES:
Percentage of union | 8 weeks post-op
Percentage of union | 12 weeks post-op
Rate of change of percent union | 8-12 weeks, 12-16 weeks
Pattern of partial union on initial CT scan | 8 weeks
Time to return to work | up to 52 weeks
Functional outcomes as measured by range of motion and grip strength | up to 52 weeks
  Range of motion measurements of wrist flexion/extension and forearm supination/pronation; grip strength using a grip dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Neil White, MD, Principal Investigator — University of Calgary
Locations (6):
- Canada (6):
  - South Health Campus, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - PanAM Clinic Foundation, Winnipeg, Manitoba
  - The Ottawa Hospital (Civic Campus), Ottawa, Ontario
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec